CLINICAL TRIAL: NCT06840678
Title: Patogénesis Cortical De La Enfermedad De Parkinson: Efectos Corticales Y Corticoestriatales De La Estimulación Transcraneal Por Campo Magnético Estático En Pacientes Con Enfermedad De Parkinson
Brief Title: Home-based Transcranial Static Magnetic Field Stimulation (tSMS) of the Supplementary Motor Area in Parkinson's Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Fundación de investigación HM (Other)
Responsible Party: Principal Investigator, Guglielmo Foffani, PhD, Fundación de investigación HM
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1715-GHM
Record Dates: First submitted 2022-12-12; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2024-04

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- tSMS (Experimental): 30 min of tSMS, 5 daily sessions per week (monday to friday), for 8 weeks, at home
  Interventions: Device: Transcranial static magnetic field stimulation (tSMS) of the supplementary motor area

INTERVENTIONS:
Device: Transcranial static magnetic field stimulation (tSMS) of the supplementary motor area — Transcranial static magnetic field stimulation (tSMS) is a non-invasive brain stimulation (NIBS) technique that decreases cortical excitability. Static magnetic fields suitable for tSMS are obtained with commercially available neodymium magnets. The investigators will use a cylindrical neodymium magnet of 60 mm diameter and 30 mm of thickness (MAG60r; Neurek SL, Toledo, Spain), which will be applied with south polarity to the supplementary motor area (SMA) using an ergonomic helmet (MAGsv1.1, Neurek SL, Toledo, Spain).
  Other Names: MAGsv1.1 with MAG60r, Neurek SL, Toledo, Spain

SUMMARY:
This is a pilot open study to test the hypothesis that home-based transcranial static magnetic field stimulation (tSMS) of the supplementary motor area is safe and feasible to modulate corticostriatal activity in patients with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* idiopathic Parkinson's disease (Brain Bank criteria)
* optimal clinical response to dopaminergic medication (>30% MDS-UPDRS-III improvement)

Exclusion Criteria:

* MRI-incompatible metal objects in the body (e.g. cardiac pacemakers)
* presence of levodopa-induced dyskinesias
* other main neuropsychiatric co-morbidity

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events (safety) | From the start to 3 months after the end of treatment (5 months)
  Number of device-related AE
Feasibility of home-based tSMS | From the start to the end of treatment (8 weeks)
  Number of home-based tSMS sessions completed, according to patient's diaries

SECONDARY OUTCOMES:
Subjective improvement | Within one week after the end of treatment compared to baseline
  Patient global impression of change (PGIC)
Motor improvement | Within one week after the end of treatment compared to baseline
  MDS-UDPRS III scale
Sleep improvement | Within one week after the end of treatment compared to baseline
  SCOPA-sleep scale

OTHER OUTCOMES:
Change in corticospinal excitability | Within one week after the end of treatment compared to baseline
  Amplitude of motor evoked potentials (MEPs) evoked by transcranial magnetic stimulation of the motor cortex
Changes in corticostriatal activity by FDG-PET | Within one week after the end of treatment compared to baseline
  FDG-PET uptake in SMA and motor striatum
Changes in corticostriatal activity by resting-state fMRI | Within one week after the end of treatment compared to baseline
  Functional connectivity between SMA and motor striatum
Changes in corticostriatal microstructure by diffusion-tensor imaging (DTI) | Within one week after the end of treatment compared to baseline
  Fractional anisotropy and diffusivity in SMA and motor striatum.

CONTACTS AND LOCATIONS:
Overall Officials: Guglielmo Foffani, PhD, Principal Investigator — HM CINAC, Hospital Universitario HM Puerta del Sur, HM Hospitales, Móstoles, Madrid, Spain
Locations (1):
- HM CINAC, Hospital Universitario HM Puerta del Sur, HM Hospitales, Móstoles, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oliviero A, Mordillo-Mateos L, Arias P, Panyavin I, Foffani G, Aguilar J. Transcranial static magnetic field stimulation of the human motor cortex. J Physiol. 2011 Oct 15;589(Pt 20):4949-58. doi: 10.1113/jphysiol.2011.211953. Epub 2011 Aug 1. PMID 21807616
- [Background] Rivadulla C, Foffani G, Oliviero A. Magnetic field strength and reproducibility of neodymium magnets useful for transcranial static magnetic field stimulation of the human cortex. Neuromodulation. 2014 Jul;17(5):438-41; discussion 441-2. doi: 10.1111/ner.12125. Epub 2013 Oct 11. PMID 24125470
- [Background] Oliviero A, Carrasco-Lopez MC, Campolo M, Perez-Borrego YA, Soto-Leon V, Gonzalez-Rosa JJ, Higuero AM, Strange BA, Abad-Rodriguez J, Foffani G. Safety Study of Transcranial Static Magnetic Field Stimulation (tSMS) of the Human Cortex. Brain Stimul. 2015 May-Jun;8(3):481-5. doi: 10.1016/j.brs.2014.12.002. Epub 2014 Dec 11. PMID 25595064
- [Background] Dileone M, Carrasco-Lopez MC, Segundo-Rodriguez JC, Mordillo-Mateos L, Lopez-Ariztegui N, Alonso-Frech F, Catalan-Alonso MJ, Obeso JA, Oliviero A, Foffani G. Dopamine-dependent changes of cortical excitability induced by transcranial static magnetic field stimulation in Parkinson's disease. Sci Rep. 2017 Jun 28;7(1):4329. doi: 10.1038/s41598-017-04254-y. PMID 28659614
- [Background] Dileone M, Mordillo-Mateos L, Oliviero A, Foffani G. Long-lasting effects of transcranial static magnetic field stimulation on motor cortex excitability. Brain Stimul. 2018 Jul-Aug;11(4):676-688. doi: 10.1016/j.brs.2018.02.005. Epub 2018 Feb 7. PMID 29500043
- [Background] Pineda-Pardo JA, Obeso I, Guida P, Dileone M, Strange BA, Obeso JA, Oliviero A, Foffani G. Static magnetic field stimulation of the supplementary motor area modulates resting-state activity and motor behavior. Commun Biol. 2019 Oct 31;2:397. doi: 10.1038/s42003-019-0643-8. eCollection 2019. PMID 31701026
- [Background] Dileone M, Ammann C, Catanzaro V, Pagge C, Piredda R, Monje MHG, Navalpotro-Gomez I, Bergareche A, Rodriguez-Oroz MC, Vela-Desojo L, Alonso-Frech F, Catalan MJ, Molina JA, Lopez-Ariztegu N, Oliviero A, Obeso JA, Foffani G. Home-based transcranial static magnetic field stimulation of the motor cortex for treating levodopa-induced dyskinesias in Parkinson's disease: A randomized controlled trial. Brain Stimul. 2022 May-Jun;15(3):857-860. doi: 10.1016/j.brs.2022.05.012. Epub 2022 May 21. No abstract available. PMID 35609815